CLINICAL TRIAL: NCT01769430
Title: Evaluating Modes of Influenza Transmission Work Package 1: Observational Study of Community Acquired Influenza
Brief Title: Evaluating Modes of Influenza Transmission Observational Study of Community Acquired Influenza
Acronym: EMIT
Status: Completed | Type: Observational
Sponsor: University of Maryland, College Park (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Donald K. Milton, Professor of Environmental Health, School of Public Health, University of Maryland, College Park
Other Study IDs: 017086-001; 1U01IP000497 (NIH); 3U01CI000446 (NIH); RC1AI086900 (NIH)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Influenza Virus Infection Transmission in Humans
Keywords: influenza virus; aerosol transmission; contact transmission; large droplet transmission; airborne infection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — viral cultures, viral RNA, viral cDNA, NP swabs, exhaled breath particles
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Community acquired respiratory infection: Measurement of exhaled breath aerosol
  Interventions: Other: Observational Study of influenza aerosol shedding -- No Intervention

INTERVENTIONS:
Other: Observational Study of influenza aerosol shedding -- No Intervention — No intervention -- observational study only

SUMMARY:
The recent swine origin influenza pandemic (2009), new emergence of swine origin H3N2v, and delayed availability of vaccine for these agents highlight the need to test and optimize public health intervention strategies to reduce transmission of influenza. We will use a new technology for biological particle collection (U.S. Provisional Patent Application No. 61/162,395, McDevitt et al., Aerosol Sci Technol 2013) to make fundamental observations on infectious respiratory droplets in a study of up to 200 naturally occurring seasonal influenza cases. We will collect respiratory droplets shed by participants while breathing normally, talking, and spontaneously coughing. We will characterize the size distribution of droplets containing infectious virus. We will use these basic data to examine the roles of large and small respiratory droplets and examine how the interaction of host factors and virus type impact the shedding of infectious respiratory droplets. Subjects will be recruited through a web based respiratory illness surveillance system, health clinics and advertisement in the campus community. Sitting in the collection booth will not create additional discomfort or risk for volunteers already suffering from influenza infection. We will recruit up to 1000 persons with symptoms of acute respiratory illness for screening with collection of nasopharyngeal swabs and questionnaire. From among those screened, we will recruit 250 to give exhaled breath samples, and ask 50 people with influenza to return for follow up exhaled breath samples on up to two subsequent days. We hypothesize that (1) fine aerosols (<5 microns in aerodynamic diameter) will contain more viral copies than coarse aerosol particles (>= 5 microns) (2) fine aerosols will contain culturable virus indicating that the fine aerosols are infectious, (3) aerosol shedding will correlate with virus load measured by swabs, (4) presence of active cough during sampling will be associated with increased aerosol shedding, (5) clinical symptoms and signs, including fever can be used to predict viral aerosol shedding.

DETAILED DESCRIPTION:
This study is a follow-on to earlier projects funded by the US Centers for Disease Control and Prevention (CDC) and the National Institute for Allergy and Infectious Diseases (NIAID) that developed the sampler and studied the impact of surgical masks on reducing viral aerosol release by persons infected with influenza virus. The funding organizations have no direct control over the study design, execution, or reporting and no access to identifiable human data. The CDC IRB has determined that the CDC is not engaged in human subjects research in this cooperative agreement.

Hypotheses:

* Fine particle aerosols will contain greater numbers of viral copies than will coarse aerosol particles.
* Clinical symptoms and signs, including fever can be used to predict viral aerosol shedding
* Fine aerosols will contain culturable virus indicating that the fine aerosols are infectious
* Aerosol shedding will correlate with virus load measured by nasopharyngeal and throat swabs
* Presence of active cough during sampling will be associated with increased aerosol shedding with a stronger correlation to be found with coarse than fine particle virus aerosols

ELIGIBILITY:
Inclusion Criteria:

* Presence of symptomatic respiratory infection or other evidence of respiratory infection:

  * During the influenza season, subjects will be enrolled if they have

    * influenza-like illness (symptoms of fever and either cough or sore throat) and either
    * a positive point of care rapid test for influenza infection or
    * objectively documented fever in the setting of a documented local influenza outbreak (presence of rapid test or PCR confirmed cases).
    * Onset within the previous 48 hours
  * Prior to onset of influenza season and if we have not achieved enrollment of our target population by the end of flu season, we will enroll subjects with cough, coryza (stuffy runny nose, sore throat, sneezing), and malaise (fatigue) characteristic of the 'common cold' often resulting from Human Rhinovirus, RSV, parainfluenza, and to some extent influenza virus.

Exclusion Criteria:

-

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Students, faculty, and staff at the University of Maryland College Park and residents of the surrounding communities
Sampling Method: Non-Probability Sample
Enrollment: 178 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald K Milton, MD, DrPH, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland School of Public Health, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The study data for natural infections are available upon request. All analysis scripts and readme files required to reproduce analyses are available at https://gitlab.com/jacob bueno /natur al_vs_ artif icial_infection
Supporting Information: SAP, Analytic Code
Time Frame: open access indefinately
Access Criteria: Open
URL: https://gitlab.com/jacobbueno/natural_vs_artificial_infection

REFERENCES:
- [Background] Fabian P, McDevitt JJ, DeHaan WH, Fung RO, Cowling BJ, Chan KH, Leung GM, Milton DK. Influenza virus in human exhaled breath: an observational study. PLoS One. 2008 Jul 16;3(7):e2691. doi: 10.1371/journal.pone.0002691. PMID 18628983
- [Background] Milton DK, Fabian MP, Cowling BJ, Grantham ML, McDevitt JJ. Influenza virus aerosols in human exhaled breath: particle size, culturability, and effect of surgical masks. PLoS Pathog. 2013 Mar;9(3):e1003205. doi: 10.1371/journal.ppat.1003205. Epub 2013 Mar 7. PMID 23505369
- [Background] McDevitt JJ, Koutrakis P, Ferguson ST, Wolfson JM, Fabian MP, Martins M, Pantelic J, Milton DK. Development and Performance Evaluation of an Exhaled-Breath Bioaerosol Collector for Influenza Virus. Aerosol Sci Technol. 2013 Jan 1;47(4):444-451. doi: 10.1080/02786826.2012.762973. Epub 2013 Jan 25. PMID 23418400
- [Result] Yan J, Grantham M, Pantelic J, Bueno de Mesquita PJ, Albert B, Liu F, Ehrman S, Milton DK; EMIT Consortium. Infectious virus in exhaled breath of symptomatic seasonal influenza cases from a college community. Proc Natl Acad Sci U S A. 2018 Jan 30;115(5):1081-1086. doi: 10.1073/pnas.1716561115. Epub 2018 Jan 18. PMID 29348203

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Self reported ILI and influenza diagnosed by campus health center
Pre-assignment Details: must have fever measured by campus medical provider or by research clinic with a sore throat or cough, or a positive rapid antigen test for influenza A or B and must be within 3 days of onset of symptoms
Groups:
- Symptomatic Influenza Virus Infection: Symptomatic influenza cases with either fever or a positive rapid antigen test.
Period: Overall Study
Arm/Group | Symptomatic Influenza Virus Infection
Started | 178 (Volunteers recruited and screened and met enrollment criteria)
Completed | 178 (Met enrollment criteria and provided samples)
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Community Acquired Influenza Virus Infection: Volunteers with positive rapid antigen test or objectively measured fever with complaint of cough or sore throat during the influenza season.
Arm/Group | Community Acquired Influenza Virus Infection
Number analyzed (Participants) | 178
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 21 [19 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 177
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 32
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 109
  More than one race | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 178

OUTCOME MEASURES:

1. Primary Outcome: Viral Copy Number in 30-minute Exhaled Breath Sample
Description: Total viral RNA copies detected in breath aerosol exhaled during a 30-minute sample collection. Participants sit for 30 minutes with face inside the cone/funnel of the Gesundheit-II (G-II) human bioaerosol collector (https://doi.org/10.1080/02786826.2012.762973) collecting air at 130 L/min. Particles in air are concentrated into a small volume of buffer. The copies per mL of buffer is measured by PCR and corrected to the total amount collected per 30-min sample. See publication in the Proceedings of the National Academy of Sciences (https://doi.org/10.1073/pnas.1716561115) and PLoS Pathogens (https://doi.org/10.1371/journal.ppat.1003205) for more details.
Time Frame: Daily measurements on days 1 through 3 post onset of symptoms (each person contributed 1 to a max of 3 samples). Reported values are the geometric mean over all samples and persons.
Population: All cases meeting enrollment criteria
Measure: Geometric Mean (Standard Deviation); unit: Fine aerosol RNA copy number
Arm/Group | Community Acquired Respiratory Infection
Number analyzed (Participants) | 178
Fine aerosol RNA copy number
  Fine aerosol RNA copy number, Total copies per 30-minute breath sample | 38,000 (13)
  Coarse aerosol RNA copy number, Total per 30-minute breath sample | 12,000 (14)

2. Primary Outcome: Total Fine Aerosol Infectious Influenza Virus in 30-minute Exhaled Breath Sample
Description: Fluorescent Focus Assay detection of infectious influenza virus in Fine Particle (≤5 µm) aerosol reported as fluorescent focus units (FFU) per 30-minute breath sample. Aerosol samples were collected at 130 L/min for 30 minutes by an aerosol sampler that concentrated the aerosol in a small volume of liquid. The FFU/ml were multiplied by the volume of liquid in the final concentrate sample to obtain the total infectious particles per 30-minute sample. This outcome was peer reviewed and published in the Proceedings of the National Academy of Sciences.
Time Frame: as for outcome 1
Population: Participants with complete data
Measure: Geometric Mean (Standard Deviation); unit: Total FFU/30-minute sample
Arm/Group | Community Acquired Respiratory Infection
Number analyzed (Participants) | 142
Total FFU/30-minute sample | 41 (30)

3. Other Pre Specified Outcome: Comparison of Exhaled Virus in Community Acquired and Experimental Infection
Description: We compared influenza A viral aerosol shedding from volunteers nasally inoculated with A/Wisconsin/2005 (H3N2) and college community adults naturally infected with influenza A/H3N2 (2012-2013), selected for influenza-like illness with objectively measured fever or a positive Quidel QuickVue A&B test. Propensity scores were used to control for differences in symptom presentation observed between experimentally and naturally infected groups.
Time Frame: Maximal shedding during days 1-3 post onset of symptoms (natural infections) or days 1-4 post inoculation (nasally inoculated volunteers)
Population: Adults naturally infected with influenza A H3N2
Measure: Geometric Mean (Standard Deviation); unit: Fine aerosol RNA copies/ 30-min sample
Groups:
- Participants Infected With Influenza A H3N2: College community adults naturally infected with influenza A/H3N2 (2012-2013), selected for influenza-like illness with objectively measured fever or a positive Quidel QuickVue A&B test from this study were compared with volunteers nasally inoculated with A/Wisconsin/2005 (H3N2) from a companion study ClinicalTrials.gov (number NCT01710111).
- Volunteers Nasally Inoculated With A/Wisconsin/2005 (H3N2): From ClinicalTrials.gov (number NCT01710111).
Arm/Group | Participants Infected With Influenza A H3N2 | Volunteers Nasally Inoculated With A/Wisconsin/2005 (H3N2)
Number analyzed (Participants) | 83 | 39
Fine aerosol RNA copies/ 30-min sample | 39000 (15.12) | 5100 (4.72)

4. Post Hoc Outcome: Correlation of Exhaled Particle Counts and Viral Copy Numbers
Description: A convenience subsample were tested for exhaled particle counts using an optical particle counter during research clinic visits as a postdoctoral exploratory investigation.
  No formal analysis was completed.
Time Frame: as for outcome 1
Population: Convenience subsample
Arm/Group | Community Acquired Respiratory Infection
Number analyzed (Participants) | 0

5. Post Hoc Outcome: Impact of Co-infection With Viral or Bacterial Pathogens on Fine Aerosol Shedding
Description: Exploratory analysis of impact of other respiratory present in nasopharyngeal swabs on extent of aerosol shedding.
Time Frame: Within 3 days of onset of influenza like illness
Population: Postdoc left lab without completing write up of analysis due to lack of finding a correlation. Notes and data from 12 years ago are no longer easily accessible.
Arm/Group | Community Acquired Respiratory Infection
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Observational Study: Symptomatic influenza cases with either fever or a positive rapid antigen test.
Arm/Group | Observational Study
All-Cause Mortality (participants affected / at risk) | 0/178
Serious Adverse Events (participants affected / at risk) | 0/178
Other Adverse Events (participants affected / at risk) | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes